CLINICAL TRIAL: NCT04420247
Title: Multicentric Pragmatic Randomized Controled Trial to Evaluate the Efficacy Chloroquine or Hydroxychloroquine for Five Days in Treating Pneumonia Caused by SARS-Cov-2 - COVID-19
Brief Title: Efficacy of Chloroquine or Hydroxychloroquine in Treating Pneumonia Caused by SARS-Cov-2 - COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro de Estudos e Pesquisa em Emergencias Medicas e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, ALVARO REA-NETO, MD, Director of the Reseach Center, Centro de Estudos e Pesquisa em Emergencias Medicas e Terapia Intensiva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOROTRIAL
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: COVID; COVID-19; SARS-CoV 2; Coronavirus; Corona Virus Infection
Keywords: VIRAL PNEUMONIA; CORONAVIRUS; COVID-19; COVID; SARS-COV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia, Viral | interventions — Chloroquine; Hydroxychloroquine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two arms - Intervention and Control Intervention received unblinded treatment with Chloroquine or Hyroxycloroquine for 5 days, as well as standard treatment available and recomended by the Brazilian Guidelines for COVID-19.
  Control group received just the standard treatment available and recomended by the Brazilian Guidelines for COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Treatment with either Chloroquine or Hydroxychloroquine according to what was available in the hospital:
  Chloroquine - 900mg on the first day, followed by 450mg in the next 4 days. Hydroxychloroquine - 800mg on the first day, followed by 450mg in the next 4 days.
  +
  Standard treatment available and recomended by the Brazilian Guidelines for COVID-19.
  Interventions: Drug: Chloroquine; Drug: Hydroxychloroquine
- Control (Active Comparator): Standard treatment available and recomended by the Brazilian Guidelines for COVID-19.
  Interventions: Other: standard care

INTERVENTIONS:
Drug: Chloroquine — 5 days of treatment with Chloroquine + Standard Care
  Arms: Intervention
Drug: Hydroxychloroquine — 5 days of treatment with Hydroxychloroquine + Standard Care
  Arms: Intervention
Other: standard care — Standard Care according to Brazilian Guidelines for treating COVID-19
  Arms: Control

SUMMARY:
Facing the challenge of finding an efficient treatment for COVID-19, the viral pneumonia caused by the Coronavirus SARS-Cov-2, this study intended to test if Chloroquine or Hydroxychloroquine, two drugs with strong in-vitro antiviral role proven by numerous studies and with a well defined safety profile established, for efficacy in treating COVID-19 and improving an ordinal primary outcome composed by a 9-levels scale, which was recomended by the World Health Organization.

DETAILED DESCRIPTION:
This is a Phase 3, Pragmatic, Multicentric Randomized Controled Trial of efficacy to test the effect of either Chloroquine or Hydroxychloroquine for 5 days in the recomended dose standardized by brazilian Ministry of Health.

Patients were randomized (1:1) using stratified randomization by hospital and severity at the moment of randomization (stipulated by use of mechanical ventilation or not) into two arms: Intervention and Control. Intervention group recieved a loading dose of 900mg of Chloroquine or 800mg of Hydroxycloroquine in the first day, followed by 450mg of chloroquine of 400mg of hydroxychloroquine. Primary and secondary outcomes were evaluated on the 5th, 7th, 10th, 14th, 28th day after randomization.

Although the outcomes presented in the latest version were updated late on ClinicalTrials.org, on October 23, 2020, these outcomes were already present in the trial protocol approved by the Brazilian National Commission for Ethics in Research on April 8, 2020 (approval number: 3960331) and amending the protocol, approved by the same National Commission on May 25, 2020 (approval number: 4044848)

ELIGIBILITY:
Inclusion Criteria:

* Adult Males and non-pregnant females that accept and sign the informed consent.
* Hospitalized with COVID-19 suspection that has collected the confirmatory test
* To have at least one of thes symptoms: Fever, coughing, throat ache or runny nose.
* To have at least one of these findings: radiological findings that indicates COVID-10 (bilatareal ground grass images); O2 saturation lower than 94% without supplementation and crackles in lung auscultation; Need of O2 supplementation; Need of Mechanical Ventilation.
* Female patients must also agree to use efficient counterceptive methods during the evaluation period.

Exclusion Criteria:

* Patients with psoriasis or other exfoliative disease, porphyria, epilepsy, myasthenia gravis, advanced liver failure or glucose-6-phosphate dehydrogenase deficiency.
* ALT / AST> 5 times the upper limit of normal.
* Severe chronic kidney disease in stage 4 or requiring dialysis (ie, eGFR <30).
* Pregnancy or breastfeeding.
* Early transfer to another hospital that is not a study site within 72 hours.
* Severe heart disease and / or a history of cardiac arrhythmia.
* Allergy to Chloroquine and / or Hydroxychloroquine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
World Health Organization (WHO) 9-levels ordinal scale (from 0-8) | 14 days after randomization
  Evaluation of the clinical status of patients on the 14th day after randomization defined by the 9-levels ordinal scale, with lower scores meaning better outcomes.

SECONDARY OUTCOMES:
World Health Organization (WHO) 9-levels ordinal scale (from 0-8) | 5, 7, 10 and 28 days after randomization
  Evaluation of the clinical status of patients on the 5th, 7th, 10th and 28th day after randomization defined by the 9-levels ordinal scale, with lower scores meaning better outcomes.
Mortality | 28 days after randomization
  All-cause mortality at 28 days after randomization
Ventilation free days | 28 days after randomization
  Number of days without need of Mechanical Ventilation at 28 days after randomization
ICU Lenght of Stay | 28 days after randomization
  ICU Lenght of Stay on survivors at 28 days after randomization
Hospital Lenght of Stay | 28 days after randomization
  Hospital Lenght of Stay on survivors at 28 days after randomization
Acute Kidney Disease incidence | 28 days after randomization
  Acute Kidney Disease incidence measured by Kidney Disease Improving Global Outcomes (KDIGO) stage 3 sometime until the 28th day after randomization.
Percentage of patients needing dialysis | 28 days after randomization
  Percentage of patients needing dialysis sometime until the 28th day.
Coagulopathy incidence | 28 days after randomization
  Presence of coagulopathy sometime until the 28th day (platelets < 150000 and/or INR >1.5 and/or KPTT > 35 seconds).
Mean of C Reactive Protein Levels | 5, 7, 10, 14 and 28 days after randomization
  Mean of C Reactive Protein Levels on the 5th, 7th, 10th, 14th and 28th day after randomization, during period of hospitalization
Sequential Organ Failure Assessment (SOFA) scores | 5, 7, 10, 14 and 28 days after randomization
  Sequential Organ Failure Assessment (SOFA) scores (range, 0-24, with higher scores indicating greater organ dysfunction) on the 5th, 7th, 10th, 14th and 28th day after randomization, during period of hospitalization.
Neutrophils/lymphocytes ratio | 5, 7, 10, 14 and 28 days after randomization
  Neutrophils/lymphocytes ratio on the 5th, 7th, 10th, 14th and 28th day after randomization, during period of hospitalization.

OTHER OUTCOMES:
Arrhythmia | 28 days after randomization
  Safety outcome: Any kind of arrhythmia identified by the attending physician at the time of the intercurrence, confirmed by an electrocardiogram (ECG), sometime until the 28th day

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Estudos e Pesquisa em Emergencias Clinicas e Terapia Intensiva, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rea-Neto A, Bernardelli RS, Camara BMD, Reese FB, Queiroga MVO, Oliveira MC. An open-label randomized controlled trial evaluating the efficacy of chloroquine/hydroxychloroquine in severe COVID-19 patients. Sci Rep. 2021 Apr 27;11(1):9023. doi: 10.1038/s41598-021-88509-9. PMID 33907251